CLINICAL TRIAL: NCT03988764
Title: Accurate Diagnosis of Diabetes for Appropriate Management
Brief Title: Monogenic Diabetes Misdiagnosed as Type 1
Acronym: ADDAM
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Constantin Polychronakos, Senior investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: ADDAM; Canscreen (Other: Research Ethics Board, MUHC)
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 1; Monogenic Diabetes; Neonatal Diabetes; Maturity-onset Diabetes in the Young (MODY); Wolfram Syndrome; Wolcott-Rallison Syndrome; Mitochondrial Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Wolfram Syndrome; Wolcott-Rallison syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and purified DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibody-negative: Patient has been found negative for at least three T1D antibodies.
  The investigators will proceed with whole exome sequencing
  Interventions: Other: None AHT
- Antibody-positive: Patient has been found to be positive for at least one T1D autoantibody.
  No further studies will be performed as part of the main study.
  Interventions: Other: None AHT

INTERVENTIONS:
Other: None AHT — No further intervention planned for either group as part of the current study.

SUMMARY:
The study has two aims:

1. To (1a) determine the frequency of monogenic diabetes misdiagnosed as type 1 diabetes (T1D) and (2) to define an algorithm for case selection.
2. To discover novel genes whose mutations cause monogenic diabetes misdiagnosed as T1D.

DETAILED DESCRIPTION:
Aim 1. The investigators will recruit 5,000 cases diagnosed as T1D under the age of 25, from 17 participating clinics across Canada. All cases will be tested for four antibodies (against proinsulin, GAD65, islet antigen 2 (IA-2), and ZnT8). Cases negative for all four will be exome-sequenced.

1. Variant annotation will be focused on known monogenic diabetes genes. Variants rated as pathogenic, likely pathogenic or of unknown significance whose zygosity fits the genetic model, will be confirmed in a clinically certified laboratory and communicated to the treating health care team. End-point is the frequency of such variants compared to their frequency in control, non-T1D exomes.
2. The following variables will be examined for the ability to predict monogenic diabetes: Negativity for all autoantibodies tested, family history, polygenic T1D risk score, age of onset, sex, glycosylated hemoglobin (HbA1c), insulin dose, and presence of syndromic features. Predictors will be analyzed by multiple regression and results subjected to jackknife (leave-one-out) validation. Machine-learning techniques may be used.

Aim 2. Variants outside known genes in non-diagnostic exomes will be annotated and examined under autosomal dominant, recessive, X-linked and mitochondrial inheritance models. Corresponding frequency cutoffs will be 0.0005, 0.01, 0.001 and 0.0005 (if heteroplasmy >70%). Formal mutation-burden analysis will be based on depth-adjusted data from the Genome Aggregation Database (gnomAD). Genes mutated in more than one unrelated proband will be examined by a statistical approach taking into account the presence of a large number of phenocopies (Akawi et al., Nat Genet. 2015;47:1363-1369). Genes that achieve statistical significance will be tested in additional cohorts with international collaborations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes under the age of 25 as either type 1 or undetermined type.

Exclusion Criteria:

* Existing T1D autoantibody testing with a positive result

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases diagnosed as type 1 diabetes or undetermined type.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of monogenic diabetes among patients diagnosed as type 1 diabetes. | 6 years
  The exomes of all patients negative for four T1D autoantibodies will be sequenced and pathogenic variants in genes known to cause monogenic diabetes will be called and annotated. The frequency of genes carrying such variants among these patients will be compared to control exomes from public databases.
Proportion of patients carrying mutations in previously unstudied genes that meet statistical criteria of pathogenicity for monogenic diabetes. | 7 years
  Exomes not found to carry a mutation (per outcome 1) will be analyzed to discover pathogenic variants in novel genes. Genes mutated in more than one unrelated probands will be statistically evaluated to see if variants in these gene occur more frequently than in control exomes. The number of probands that is needed to fulfill this criterion will depend on the gene's tolerance to protein-altering mutations.

SECONDARY OUTCOMES:
Risk-prediction score for monogenic diabetes mutation in antibody negative T1D patients | 5 years
  Composit score with a statistically significant ROC curve for predicting monogenic diabetes in individuals previously diagnosed as T1D. It will be based on age of onset, T1D polygenic risk score. The risk score will aim to predict monogenic diabetes in cases with clinical T1D diagnosis and known to be antibody negative. The scale will be calculated as follows: From the exome sequencing, the investigators will be able to determine genotype at the three most important loci determining risk for autoimmune T1D (HLA, INS and PTPN22).The composite risk score, along with family history, age of onset, HbA1c+4*insulin dose/kg (as proxy for residual beta cell function) will be subjected to logistic regression for an overall risk. The ROC curve will be used to select a point likely to capture most cases unlikely to have autoimmune T1D, sacrificing specificity to maximize sensitivity. Data will be validated with jackknife cross-validation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized exome data will be deposited in publicly available databases.15
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 15 years
Access Criteria: Approval, by the sponsor, of a research plan that proposes to use the data to promote diabetes research